CLINICAL TRIAL: NCT00341562
Title: Genomics of In-Stent Restenosis: Endarterectomy Study
Brief Title: Genomics of In-Stent Restenosis
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999905234; 05-H-N234
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2006-07

CONDITIONS: In-Stent Restenosis; Vascular Disease
Keywords: Gene Expression Profiling; Vascular Disease
MeSH Terms: conditions — Vascular Diseases

SUMMARY:
This study, conducted in Argentina at the Hospital Espa ol de la Plata and the Hospital Franc s de Buenos Aires, in collaboration with the NHLBI, will investigate possible genetic factors that lead to in-stent restenosis. A stent is a wire mesh tube that is surgically placed to open a blocked artery. The stent stays in the artery permanently, holding it open to improve blood flow. In the case of blocked coronary arteries, the stent improves blood flow to the heart muscle, relieving symptoms such as chest pain and shortness of breath. Sometimes re-growth of tissue within a stent, called in-stent restenosis, leads to narrowing of the artery, decreased blood flow, and a recurrence of symptoms. Genetic analysis may allow the identification of patient that may be at increased risk for in-stent restenosis and lead to methods of prevention and treatment.

Patients 18 years of age and older who are undergoing coronary endarterectomy (surgery to remove plaque from an artery) to treat in-stent restenosis at the Hospital Espa ol de la Plata and the Hospital Franc s de Buenos Aires may be eligible for this study.

Participants will have a blood sample drawn and undergo coronary endarterectomy. Tissue removed from the patient's artery or the stent during surgery will be analyzed for gene expression profiling and genotyping. The results will be studied along with information about the patients' medical history.

DETAILED DESCRIPTION:
Our laboratory is investigating the genetic basis of the vascular disease, in-stent restenosis. We hypothesize that patients with in-stent restenosis have abnormal expression of cell cycle regulatory and inflammatory genes that lead to accelerated development of vascular lesions following angioplasty, and that there is a genetic component underlying individual differences to vascular injury. We are conducting an investigation of human subjects with in-stent restenosis, entitled the CardioGene Study. The objective of the CardioGene study is to identify the genetic profile of patients at risk for in-stent restenosis. The CardioGene study completed enrollment of 465 patients in December 2004. Analysis of blood gene expression profiles, proteomic and genotyping data is currently ongoing. All analyses are conducted using peripheral blood. Concurrent analysis of restenosis tissue samples would be valuable in defining the molecular genetics of the disease.

In this complementary study of endartectomy tissues, we will collect diseased restenosis tissues removed from patients as part of their routine clinical care. We will also collect blood at the time of tissue harvesting for genomic analysis, in addition to clinical data. Genomic data will be compared to the CardioGene study findings, for the purposes of validation as well as more detailed understanding of the biology of restenosis, by investigation the molecular mechanisms of restenosis in the tissue samples.

ELIGIBILITY:
* INCLUSION CRITERIA

Patients 18 years of age or older

Patients undergoing coronary endarterectomy as part of their course of medical therapy. The lesion for which endarterectomy is being performed is restenosis within a bare metal stent within a native coronary artery

EXCLUSION CRITERIA

Current enrollment in a clinical trial for the treatment or prevention of in-stent restenosis.

Lesion within saphenous vein graft following coronary artery bypass grafting

Patients younger than 18 years of age

The patient is unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2005-09; Study Completion 2006-07

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Hayashi S, Watanabe N, Nakazawa K, Suzuki J, Tsushima K, Tamatani T, Sakamoto S, Isobe M. Roles of P-selectin in inflammation, neointimal formation, and vascular remodeling in balloon-injured rat carotid arteries. Circulation. 2000 Oct 3;102(14):1710-7. doi: 10.1161/01.cir.102.14.1710. PMID 11015352